CLINICAL TRIAL: NCT02442414
Title: A Phase 1 Study of KBP-5209 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sihuan Pharmaceutical Holdings Group Ltd. (Industry)
Collaborators: Covance (Industry); XuanZhu Pharma Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5209-CPK-1001
Record Dates: First submitted 2015-04-29; First posted 2015-05-13 (Estimated); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Advanced Solid Tumors
Keywords: Cancer; Advanced Solid Tumors; EGFR; HER2; HER3; HER4; ALK mutations; irreversible tyrosine kinase inhibitor; Metastatic Non Small Cell Lung Cancer; Gastric Cancer; Colorectal Cancer
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung; Stomach Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- KBP-5209 (Experimental): Dose escalation for KBP-5209 will initially follow a modified accelerated titration design with a starting dose of 20 mg QD. Early dose escalation will proceed with one-patient cohorts and 100% dose increments (ie, dose doubling) until a patient experiences a DLT, at which point the cohorts will move to a 3+3 design. Treatment will continue until there appears evidence of progressive disease, intolerable toxicity, or the subject discontinues from the study treatment for other reasons. A cycle is defined as continuous treatment for 28 days.
  Interventions: Drug: KBP-5209

INTERVENTIONS:
Drug: KBP-5209 — Single oral dose beginning at 20 mg with daily dosing for 28 day cycles.

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose of KBP-5209 as a single agent when given orally to adult patients with advanced solid tumors that have progressed despite standard therapy, or where there is no standard therapy.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, multicenter study of KBP-5209 administered orally once daily (QD) in 28-day treatment cycles to adult patients with advanced solid tumors which have progressed despite standard therapy or for which no standard therapy exists. This study is designed to determine the MTD or RP2D and to characterize the safety, tolerability, and PK profile of KBP-5209.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older;
* Patients with histologically or cytologically confirmed, advanced solid tumors which have progressed despite standard therapy or for whom no standard therapy exists.
* Patients must have at least one measurable or non-measurable lesion (dose escalation only) as defined by RECIST v1.1
* Eastern Cooperative Oncology Group performance score 0 to 2;

Exclusion Criteria:

* Patients with symptomatic CNS metastases;
* Patients who have a known history of hepatitis C or chronic active hepatitis B or a known diagnosis of HIV
* Any significant ophthalmologic abnormality
* Patients who have any severe and/or uncontrolled medical conditions
* Significant gastrointestinal abnormalities,
* Patients who have impaired cardiac function or clinically significant cardiac diseases,
* Chemotherapy, biologic therapy, immunotherapy, radiotherapy or investigational agents within 5 half-lives or within 4 weeks (whichever is longer) prior to administration of the first dose of study drug on Day 1 or have not recovered from the side effects of such therapy;
* Treatment with third generation EGFR inhibitors
* Major surgery/surgical therapy for any cause within 4 weeks of Screening;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-04-07 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
Outcome Measure: safety and tolerability, based on the rate of dose-limiting toxicities, toxicity grade, and reversibility of toxicity. | 2 Years

SECONDARY OUTCOMES:
Dose-dependency of toxicity based on: dose limiting toxicities; frequency, type, grade, and seriousness, and causality of treatment-emergent adverse events, and laboratory assessments. | While undergoing study treatment and up to 30 days after the last dose of KBP-5209

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah

REFERENCES:
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Simon R, Freidlin B, Rubinstein L, Arbuck SG, Collins J, Christian MC. Accelerated titration designs for phase I clinical trials in oncology. J Natl Cancer Inst. 1997 Aug 6;89(15):1138-47. doi: 10.1093/jnci/89.15.1138. PMID 9262252
- [Background] Gibaldi M, Perrier D. Pharmacokinetics. 2nd edition. New York, NY: Marcel Dekker, Inc.; 1982.
- [Background] ICH E3: Guideline for Industry: Structure and Content of Clinical Study Reports. 1996.
- [Background] Jaiswal BS, Kljavin NM, Stawiski EW, Chan E, Parikh C, Durinck S, Chaudhuri S, Pujara K, Guillory J, Edgar KA, Janakiraman V, Scholz RP, Bowman KK, Lorenzo M, Li H, Wu J, Yuan W, Peters BA, Kan Z, Stinson J, Mak M, Modrusan Z, Eigenbrot C, Firestein R, Stern HM, Rajalingam K, Schaefer G, Merchant MA, Sliwkowski MX, de Sauvage FJ, Seshagiri S. Oncogenic ERBB3 mutations in human cancers. Cancer Cell. 2013 May 13;23(5):603-17. doi: 10.1016/j.ccr.2013.04.012. PMID 23680147
- [Derived] Li M, Liu F, Zhang F, Zhou W, Jiang X, Yang Y, Qu K, Wang Y, Ma Q, Wang T, Bai L, Wang Z, Song X, Zhu Y, Yuan R, Gao Y, Liu Y, Jin Y, Li H, Xiang S, Ye Y, Zhang Y, Jiang L, Hu Y, Hao Y, Lu W, Chen S, Gu J, Zhou J, Gong W, Zhang Y, Wang X, Liu X, Liu C, Liu H, Liu Y, Liu Y. Genomic ERBB2/ERBB3 mutations promote PD-L1-mediated immune escape in gallbladder cancer: a whole-exome sequencing analysis. Gut. 2019 Jun;68(6):1024-1033. doi: 10.1136/gutjnl-2018-316039. Epub 2018 Jun 28. PMID 29954840